CLINICAL TRIAL: NCT04021563
Title: A Phase I Study to Evaluate the Safety, Tolerability, Pharmacokinetics of SR419 in Healthy Volunteers
Brief Title: The Safety, Tolerability, Pharmacokinetics(PK) of SR419 in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Shanghai SIMR Biotechnology Co., Ltd. (Industry)
Collaborators: Syneos Health (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Treatment
Other Study IDs: SR419-101
Record Dates: First submitted 2019-07-09; First posted 2019-07-16 (Actual); Last update posted 2024-11-29 (Actual); Status verified 2024-11

CONDITIONS: Healthy Volunteers

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- SR419 (Experimental): Ascending single and multiple doses of SR419 orally
  Interventions: Drug: SR419
- Placebo (Placebo Comparator): Ascending single and multiple doses of placebo orally
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: SR419 — Ascending single and multiple doses of SR419 orally
  Arms: SR419
Drug: Placebo — Ascending single and multiple doses of placebo orally
  Arms: Placebo

SUMMARY:
This study is to evaluate the safety, tolerability, PK of SR419 in healthy volunteers.

DETAILED DESCRIPTION:
This is a Phase I study to evaluate the safety, tolerability, PK of SR419 in healthy volunteers. The study will include 3 parts.

Part A is a double-blind, randomized, placebo-controlled, single-dose escalation study of SR419 in healthy young subjects.

Part B is a double-blind, randomized, placebo-controlled, repeated-dose escalation study of SR419 in healthy young subjects.

Part C is a double-blind, randomized, placebo-controlled, repeated dose study of SR419 in healthy elderly subjects.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy males and females who are 18 to 64 years of age inclusive are eligible for Parts A and B.
2. Healthy males and females who are 65 to 80 years of age inclusive, defined as elderly subjects in this study, are eligible for Part C only.
3. Average of triplicate QTcF values must be < 450 msec for males and < 470 msec for females at Screening and Day -1.
4. Bodyweight > 50 kg (110 pounds) and body mass index (BMI) between 18 and 30 kg/m2
5. The participants must agree to use contraception methods (outlined in Appendix 1)
6. Capable of giving written informed consent, which includes compliance with the requirements and restrictions listed in the consent form.
7. Male subjects must agree to use contraception methods (outlined in Appendix 1) if they have a female partner of childbearing potential and must agree not to donate sperm. This criterion must be followed from the time of the first dose of investigational medicinal product (IMP) until at least 90 days after the last dose of IMP. This requirement does not apply to subjects in a same-sex relationship and female partners of non-childbearing potential.
8. A female subject is eligible to participate if she is:

   a. of non-childbearing potential, defined as: i. Pre- menopausal females with a documented tubal ligation, tubal occlusion procedure followed by a hysterosalpingogram that confirmed bilateral tubal occlusion, bilateral salpingectomy, hysterectomy or other documented medical conditions which cause infertility and are considered to be of non-childbearing potential; ii. Postmenopausal defined as 12 months of spontaneous amenorrhea (in questionable cases a blood sample with follicle stimulating hormone [FSH] >40 mIU/mL is confirmatory). b. of childbearing potential, and one of the following applies: i. Is willing to practice true abstinent from the time of consent until at least 30 days after the last dose of IMP or 5× half-lives of the IMP, whichever is longer; ii. Agrees to comply with the protocol defined contraception requirements outlined in Appendix 1 from at least 1 month before her first dose of IMP, and until at least 30 days after her last dose of IMP or 5× half-lives of the IMP, whichever is longer.
9. Capable of giving written informed consent, which includes compliance with the requirements and restrictions listed in the consent form.

Exclusion Criteria:

1. Clinically significant history of central nervous system (CNS) disease, such as cognitive disorder and seizures. History of non-clinically significant mild anxiety (related to social stressors) or situational sleep disturbance > 6 months ago could be enrolled under the discretion of the Investigators.
2. Known history of renal dysfunction or creatinine clearance < 90 mL/min or ≥ 150 mL/min (calculated using the Cockcroft-Gault formula) at Screening.
3. Current or chronic history of liver disease or known hepatic or biliary abnormalities (with the exception of Gilbert's syndrome [indirect bilirubin < 5 mg/dL with no other clinically significant abnormalities seen] or asymptomatic gallstones).
4. History of regular alcohol consumption within 6 months of screening defined as: an average weekly intake of >21 units for males or >14 units for females. One unit is equivalent to 8 g of alcohol: a half-pint (~285 mL) of beer, 1 glass (125 mL) of wine or 1 measure (25 mL) of spirits.
5. History of significant drug abuse within one year of screening or use of soft drugs (such as marijuana) within 3 months prior to screening or hard drugs (such as cocaine, methamphetamine, crack) within 1 year prior to screening.
6. History of sensitivity to any of the IMPs, or components thereof or a history of drug or other allergy that, in the opinion of the Investigator or Medical Monitor, contraindicates participation.
7. History of asthma (excluding resolved childhood asthma), anaphylaxis or anaphylactoid reactions, severe allergic responses.
8. History of hypercoagulable state or history of thrombosis.
9. A history of biliary tract disease including a history of liver disease with elevated liver function tests of known or unknown etiology (with the exception of Gilbert's syndrome).
10. A positive pre-study Hepatitis B surface antigen or positive Hepatitis C antibody result within 3 months of screening.
11. Use of tobacco- or nicotine-containing products:

    1. Parts A and B: positive urinary cotinine test at Screening or Day -1 or history of regular use of tobacco- or nicotine-containing products (more than 4 products per month within 6 months prior to screening) or unwilling to refrain from use of such products from Screening until completion of the final study visit;
    2. Part C: positive urinary cotinine test at Screening or Day -1 or history of regular use of tobacco- or nicotine-containing products (more than 4 products per month within 6 months prior to screening) or unwilling to give up these products from Screening until discharge from the study unit.
12. A positive pre-study drug/alcohol result at Screening or Day -1.
13. A positive test for human immunodeficiency virus (HIV) antibody.
14. Donation or lost in excess of 500 mL of blood within 56 days of Day 1 or donation of plasma within 14 days of Day 1.
15. The subject has participated in a clinical trial and has received an investigational product within the following time period prior to the first dosing day in the current study: 30 days, 5 half-lives or twice the duration of the biological effect of the investigational product (whichever is longer).
16. Exposure to more than four new chemical entities within 12 months prior to the first dosing day.
17. Use of medication other than topical products without significant systemic absorption:

    1. prescription within 14 days and over-the-counter (OTC) medications within 7 days, or 5× half-lives (whichever is longer) prior to the first dose of IMP, with the exception of the occasional use of paracetamol (up to 2 g daily)
    2. natural health products (e.g. food supplements and herbal supplements) within 7 days prior to the first dose of IMP;
    3. a depot injection or an implant of any drug within 3 months prior to the first dose of IMP.
    4. vaccine within 1 month prior to the first dose of IMP.
18. Unable to refrain from consumption of Seville oranges, grapefruit or grapefruit juice within 7 days prior to the first dose of IMP until the Safety Follow-up visit.
19. A positive pre-study pregnancy test at Screening or Day -1.
20. Breast-feeding and/or lactating subject.
21. Any reason which, in the opinion of the Investigator, would prevent the subject from participating in the study.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2019-07-26 (Actual); Primary Completion 2019-12-10 (Actual); Study Completion 2019-12-10 (Actual)

PRIMARY OUTCOMES:
The frequency and severity of AEs in healthy volunteers adminstrated with single and repeated oral doses of SR419 | Up to Day14 for the safety follow up since Day1
  AE: adverse event
Heart rate changes since baseline (categorized as normal; abnormal, not clinically significant; and abnormal, clinically significant) | Up to Day14 for the safety follow up since Day1
PR interval changes since baseline (categorized as normal; abnormal, not clinically significant; and abnormal, clinically significant) | Up to Day14 for the safety follow up since Day1
QRS duration changes since baseline (categorized as normal; abnormal, not clinically significant; and abnormal, clinically significant) | Up to Day14 for the safety follow up since Day1
QT interval changes since baseline (categorized as normal; abnormal, not clinically significant; and abnormal, clinically significant) | Up to Day14 for the safety follow up since Day1
QTcF changes since baseline (categorized as normal; abnormal, not clinically significant; and abnormal, clinically significant) | Up to Day14 for the safety follow up since Day1
Systolic blood pressure changes since baseline | Up to Day14 for the safety follow up since Day1
Diastolic blood pressure changes since baseline | Up to Day14 for the safety follow up since Day1
Pulse rate changes since baseline | Up to Day14 for the safety follow up since Day1
Respiratory rate changes since baseline | Up to Day14 for the safety follow up since Day1
Oral temperature changes since baseline | Up to Day14 for the safety follow up since Day1

SECONDARY OUTCOMES:
Cmax | Up to Day 9
  Peak plasma concentration
Tmax | Up to Day 9
  Time of peak plasma concentration
AUC | Up to Day 9
  Area under the plasma concentration-time curve
CL/F | Up to Day 9
  Apparent total clearance
t1/2 | Up to Day 9
  Terminal half-life
R0 | Up to Day 9
  Accumulation ratio
Ae | Up to Day 9
  The amount of drug excreted unchanged in the urine
CLr | Up to Day 9
  Renal clearance

CONTACTS AND LOCATIONS:
Overall Officials: Dr.Hatchuel, Principal Investigator — Linear Clinical Research
Locations (1):
- Linear Clinical Research, Perth, Australia

IPD SHARING:
Plan to Share IPD: No